CLINICAL TRIAL: NCT01336374
Title: A Pilot Randomized Controlled Trial of Vacant Lot Greening and Violence-related Outcomes
Brief Title: Vacant Lot Greening and Violence-Related Outcomes
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 813112
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Violence Prevention; Built Environment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Greened Vacant Lot: A cluster of vacant lots is greened. People living around this area make up this cohort.
- Control Site: The control site is a cluster of vacant lots that will not be greened. The people living around these lots make up the control group.

SUMMARY:
The purpose of this study is to determine the impact of vacant lot greening on perceptions of safety and violence for residents living around the lots. We hypothesize that people living around lots that are greened will have improved perception of safety.

DETAILED DESCRIPTION:
Violence is a serious health problem in the US, and especially in Philadelphia, as the city ranks first in violent crime amongst the ten largest US cities. The determinants of violent crime range from individual to community level factors. In this study, we focus on physical incivilities in the built environment, specifically vacant lots, as they have been associated with violent crime. Physical incivilities are also associated with individual perceptions of crime and safety, and subsequently, negative health outcomes. However, prior research has been observational and retrospective. We aim to expand this body of work through a randomized community intervention trial of vacant lot greening to explore causal mechanisms between vacant lots and violent crime outcomes. This pilot study, in partnership with the Pennsylvania Horticultural Society, will investigate the feasibility of a vacant lot greening intervention, and explore how vacant lot greening changes resident perception about violence, fear, stress, and neighborhood disorder, as well as violent crime in the surrounding area. We will interview residents living around the greened and non-greened lots during a joint walk around a pre-determined route, which will ensure exposure to our intervention. We will also use violent crime data (homicide, aggravated assault, robbery, and rape) from the Philadelphia Police Department. Results of this pilot trial will be used to develop a full scale vacant lot greening grant to be submitted to the National Institutes of Health or the National Institute of Justice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Lives in home
* Ability to walk unassisted and without difficulty for 10 blocks

Exclusion Criteria:

* One resident per house

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents living around two seperate sites (one site where vacant lots are greened and a control site where vacant lots are not greened).
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Perceptions of safety and violence | measured twice - once during first month of study and once during 4th or 5th month.
  We will be performing qualitative interviews to assess perceptions of safety and violence. We will compare these perceptions over time between two groups.

SECONDARY OUTCOMES:
Heart Rate | measured twice - once during first month of study and once during 4th or 5th month of study
  Participants wear a heart rate monitor during a walk around their neighborhood.
Violent crime statistics | Measured 6 months before intervention and 6 months after intervention
  We will obtain crime statistics, including homicide, robbery, rape, and assault in the area around each cluster of vacant lots.
Safe/Unsafe items in the environment | measured twice - once during the first month of the study and once during the 4th or 5th month.
  During a walk around the neighborhood, participants will point out items in the environment which they feel are safe or unsafe.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia C Garvin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States